CLINICAL TRIAL: NCT04909788
Title: Factors and Characteristics of Heart Rate Variability During Long Distance Running
Brief Title: Factors and Characteristics of Heart Rate Variability in Runners
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Sheng Wei, professor, Huazhong University of Science and Technology
Other Study IDs: 2021-S039
Record Dates: First submitted 2021-05-26; First posted 2021-06-02 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Heart Rate Variability; Sports Accident

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults with regular exercise: Subjects will be asked to wear a small monitoring equipment before,during and after a long distance running (over 3 km).
  Interventions: Behavioral: a long-distance running (over 3 km)

INTERVENTIONS:
Behavioral: a long-distance running (over 3 km) — Complete a long distance running（over 3 km） within the specified time (30 minutes)

SUMMARY:
The purpose of this study is to describe the variation characteristics and factors of the heart rate variability during long-distance running.

DETAILED DESCRIPTION:
Heart rate variability is recognized as the indicator to measure the autonomic nerve activity. By monitoring the heart rate variability of runners during long-distance running, we could monitor the status of the runners' cardiovascular system and predict the exercise risk of runners during long-distance running.

ELIGIBILITY:
Inclusion Criteria:

People have below conditions could be included:

1. age is 18-60 years.
2. have normal ECG .
3. agree to participate in the study.

Exclusion Criteria:

People have below conditions will be excluded:

1. have known Congenital heart disease and rheumatic heart disease.
2. have known Hypertension and cerebrovascular disease.
3. have known Myocarditis and other heart diseases.
4. have known Coronary artery disease and severe arrhythmia.
5. have known Diabetes with high or low blood glucose.
6. have a cold within two weeks before the study.
7. have other diseases considered unsuitable for participants in this study.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults with regular exercise
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
change of heart rate variability | up to 1 year
  Subjects will be asked to wear a small monitoring equipment before,during and after a long distance running (over 3 km)， and complete the corresponding amount of exercise within a specified time during the test

CONTACTS AND LOCATIONS:
Overall Officials: sheng wei, professor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Zhou Qin, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hua W, Zhang LF, Wu YF, Liu XQ, Guo DS, Zhou HL, Gou ZP, Zhao LC, Niu HX, Chen KP, Mai JZ, Chu LN, Zhang S. Incidence of sudden cardiac death in China: analysis of 4 regional populations. J Am Coll Cardiol. 2009 Sep 15;54(12):1110-8. doi: 10.1016/j.jacc.2009.06.016. No abstract available. PMID 19744622
- [Background] Iskandar EG, Thompson PD. Exercise-related sudden death due to an unusual coronary artery anomaly. Med Sci Sports Exerc. 2004 Feb;36(2):180-2. doi: 10.1249/01.MSS.0000113685.89906.04. PMID 14767237